CLINICAL TRIAL: NCT05560126
Title: Validation of the Canadian Prehospital Syncope Risk Score
Brief Title: Canadian Prehospital Syncope Risk Score (Prehospital CSRS)
Status: Not yet recruiting | Type: Observational
Sponsor: Venkatesh Thiruganasambandamoorthy (Other)
Responsible Party: Sponsor-Investigator, Venkatesh Thiruganasambandamoorthy, Principal Investigator, Ottawa Hospital Research Institute
Organization: Ottawa Hospital Research Institute (Other)
Other Study IDs: 4136
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-03

CONDITIONS: Syncope
Keywords: Syncope; Emergency Medicine Services; Prehospital; Risk-stratification; Emergency Department
MeSH Terms: conditions — Syncope; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background: Syncope is defined as a sudden, brief loss of consciousness (LOC) followed by a rapid complete recovery. It accounts for 160,000 emergency department (ED) visits each year in Canada. Despite this, few people are hospitalized (~15%) and even fewer will die (~1%). Two-thirds of patients with syncope arrive at the ED by calling 911. There are many causes of syncope. Identifying patients at low risk for bad outcomes would allow paramedics to safely determine which patients need care in the ED from those who can remain home. The research team recently developed the Canadian Prehospital Syncope Risk Score (CPSRS) which accurately identified patients at low risk for 30-day serious outcomes.

Objective: The goal of this study is to validate the accuracy of the CPSRS in the prehospital setting or refine if needed to predict the risk of 30-day serious outcomes for patients with syncope.

Methods: The research team will enroll patients with syncope from five paramedic services across Canada (British Columbia - Vancouver and Kelowna areas only, London-Middlesex, York Region, Frontenac, and Ottawa). The research team will exclude patients <18 years old, LOC >5 minutes, changes in mental status from baseline, alcohol or drug intoxication, or language barrier. Paramedics will fill out a study data collection form with the CPSRS items and additional data should the tool need refinement. The data will be entered into a secure database and will assess patient outcomes (death and potentially life-threatening medical conditions) at 30 days. The research team will examine model accuracy using standard prediction measures and look to improve model accuracy if needed. The research team expects to enroll 4875 patients over a 1-year recruitment period based on annual call volumes.

Expected Outcomes: Once validated, the tool could reduce the number of patients transported to the hospital by identifying those at low risk. This would improve patient-oriented care, while at the same time saving valuable paramedic and ED resources.

DETAILED DESCRIPTION:
The study will include patients from British Columbia (BC) Emergency Health Services (Vancouver and Kelowna areas only), London-Middlesex Paramedic Services - receiving hospitals: London Health Science Centre, York Region Paramedic Services - receiving hospital Markham Stouffville Hospital, Southlake Regional Health Centre, Mackenzie Health (Richmond Hill and Vaughan Hospital), Frontenac Paramedic Services - receiving hospitals: Kingston General Hospital, Hotel Dieu Hospital, and Ottawa Paramedic Services - receiving hospitals: The Ottawa Hospital (Civic and General campus), Queensway Carleton Hospital, Montfort Hospital.

Consecutive 911 patients will be screened by paramedics during their initial assessment. Patients meeting the above inclusion and exclusion criteria will be enrolled in the study. The research team will collect data for the CPSRS validation as well as additional variables for tool refinement if necessary. The additional variables were identified through literature, and experts in areas of syncope, prehospital, and emergency medicine. The research team will prospectively collect data in the prehospital setting, and through records review in both prehospital and in-hospital settings.

The research team will assess for outcome occurrence using a stepwise approach: 1) Review of prehospital records including ECG; 2) ED and inpatient hospital records during the index ED or any return ED visits including autopsy records for those who died, outpatient clinical notes and results of outpatient investigations available in the electronic medical records. 3) The research team will conduct a 30-day outcome assessment by telephone follow-up to verify that the patient is alive and has not sustained any SAE. During follow-up, The research team will ask questions regarding ED or outpatient clinic visits after the index event, any new diagnosis or procedural interventions, and if the cause for the syncope has been identified. The questions will require a yes/no answer. If the patient has difficulty comprehending the questions, the research team will assist the patient to understand the meaning of the questions. In addition to the questions for outcome assessment, the research team will ask patients their comfort with paramedics using the CPSRS to make disposition decisions. Our team has successfully used similar follow-up for outcomes in previous clinical decision rule studies. The research team will also work with Institute for Clinical Evaluative Sciences (ICES) or Population Data BC to check for deaths, return to ED, hospitalization, and device insertion for 1-year outcomes. Final determination of SAE will be completed by an independent Adjudication Committee blinded to the predictor variables comprised of three investigators (1 advanced care paramedic and 2 ED physicians).

The research team plans to complete the study over a twenty-one-month period which is highly feasible. The first three months are for study preparation, 12 months of data collection, and 3 months for data cleaning and analysis. The research team will publish and undertake end-of-grant knowledge translation (KT) activities during the last three months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who access paramedic services through the 911 system will be included if they have suffered syncope, defined as a sudden transient loss of consciousness followed by spontaneous complete recovery.

Exclusion Criteria:

* Pediatric patients (<18 years old),
* Patients who have a prolonged period of unconsciousness (>5 minutes),
* Change in mental status from baseline, witnessed seizure,
* Loss of consciousness due to head trauma (i.e., trauma was the initial event),
* or if unable to provide accurate details due to language barrier, cognitive impairment, alcohol, or drug intoxication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who access paramedic services through the 911 system will be included if they have suffered syncope, defined as a sudden transient loss of consciousness followed by spontaneous complete recovery.
Sampling Method: Non-Probability Sample
Enrollment: 4875 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
A serious adverse event (SAE) occurring within 30 days of the 911 call | 30 days after the 911 call
  The definition of SAE is consistent with our previous syncope research studies including the CPSRS derivation and comprises of any one of the following: a) Death due to a cause of syncope or an unknown cause; b) Arrhythmia; c) Myocardial infarction; d) Identification of serious structural heart disease; e) Aortic dissection; f) Pulmonary embolism; g) Severe pulmonary artery hypertension; h) Subarachnoid hemorrhage; i) Significant hemorrhage; j) Other serious conditions such as ectopic pregnancy, pneumothorax, or sepsis that will require treatment, or any intervention used to treat a cause of syncope.

CONTACTS AND LOCATIONS:
Overall Officials: Venkatesh Thiruganasambandamoorthy, CCFP-EM, MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We don't have no plan to share IPD